CLINICAL TRIAL: NCT04382053
Title: Phase 2, Randomized, Controlled, Open Label Multi-center Study to Assess Efficacy and Safety of DFV890 for the Treatment of SARS-CoV-2 Infected Patients With COVID-19 Pneumonia and Impaired Respiratory Function
Brief Title: Study of Efficacy and Safety of DV890 in Patients With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDFV890D12201; 2020-001870-32 (EudraCT Number)
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-06

CONDITIONS: COVID-19 Pneumonia, Impaired Respiratory Function
Keywords: COVID-19 pneumonia; SARS-CoV-2; APACHE II; DFV890; inflammasome
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DFV890 + SoC (Experimental): DFV890 50 mg was administered orally or nasogastrically twice per day (b.i.d) approximately 12 hours apart (morning and evening) for 14 days in addition to SoC.
  Interventions: Drug: DFV890; Drug: Standard of Care (SoC)
- Standard of Care (SoC) (Active Comparator): SoC was used as an active comparator arm.
  Interventions: Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: DFV890 — DFV890 25 mg tablets orally/nasogastrically administered 50 mg b.i.d for 14 days in addition to SoC.
  Arms: DFV890 + SoC
Drug: Standard of Care (SoC) — SoC included a variety of supportive therapies that ranged from the administration of supplementary oxygen to full intensive care support, alongside the use of antiviral treatment, convalescent plasma, corticosteroids, antibiotics or other agents.

SUMMARY:
This clinical study was designed to assess the efficacy and safety of DFV890 for the treatment of severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2) infected patients with coronavirus disease 2019 (COVID-19) pneumonia and impaired respiratory function.

DETAILED DESCRIPTION:
This was a Phase II, randomized, controlled, open label multi-center study to assess the efficacy and safety of DFV890 for the treatment of SARS-CoV-2 infected patients with COVID-19 pneumonia and impaired respiratory function.

The study consisted of four distinct study periods:

Screening / Baseline visit (Day -1 to 1): lasted up to a maximum of 24 hours and comprised a screening / baseline assessment. This visit was used to confirm that the study inclusion and exclusion criteria were met and served as baseline assessment prior to randomization.

Treatment period (Day 1-15): Participants were randomized as soon as possible, but within a maximum of 24 hours after screening in a 1:1 ratio receiving either DFV890 in addition to standard of care (SoC) or SoC alone. Participants in the investigational treatment arm received DFV890 administered for a total of 14 days in addition to SoC. Participants in the control arm received SoC alone. Study assessments were conducted every 2 days for hospitalized participants.

The End of Treatment (EOT) visit took place on Day 15. If participants were discharged from the hospital prior to Day 15, assessments on the day of discharge were performed according to the schedule listed under Day 15; participants continued to take the investigational treatment at home to complete the 14-day treatment period and the participants returned to the site for the Day 15/EOT assessment. If a hospital visit was not possible at Day 15, then home nursing services were used to support the last visit.

Follow-up (Day 16-29): After completion of the treatment period, participants were observed until Day 29 or discharged from hospital, whichever was sooner. Study assessments were conducted every 2 days for hospitalized participants. If participants were discharged from hospital prior to Day 29, a study visit conducted by telephone was performed on Day 29.

30-day safety follow-up assessment (Day 45): A follow-up visit for safety was conducted by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-80 years inclusive at screening.
* Clinically diagnosed with the SARS-CoV-2 virus by polymerase chain reaction (PCR) or by other approved diagnostic methodology within 7 days prior to randomization.
* Hospitalized with COVID-19-induced pneumonia evidenced by chest X-ray, computed tomography scan (CT scan) or magnetic resonance scan (MR scan), taken within 5 days prior to randomization (within 24 hours in patients in the Netherlands).
* Impaired respiratory function, defined as peripheral oxygen saturation (SpO2) ≤93% on room air or partial pressure of oxygen (PaO2) / fraction of inspired oxygen (FiO2) <300 millimeter of mercury (mmHg) at screening. For cities located at altitudes greater than 2500 m above sea level, these will be substituted with SpO2 <90% and PaO2/FiO2 <250 mmHg.
* APACHE II score of ≥10 at screening.
* C-reactive protein (CRP) ≥20 mg/L and/or ferritin level ≥600 μg/L at screening.
* Body mass index of ≥18 to <40kg/m2 at screening.

Exclusion Criteria:

* Suspected active or chronic bacterial (including Mycobacterium tuberculosis), fungal, viral, or other infection (besides SARS-CoV-2).
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatment.
* Intubated prior to randomization.
* Previous treatment with anti-rejection and immunomodulatory drugs within the past 2 weeks, or within the past 30 days or 5 half-lives (whichever is the longer) for immunomodulatory therapeutic antibodies or prohibited drugs, with the exception of hydroxychloroquine, chloroquine or corticosteroids:

For COVID-19 infection, ongoing corticosteroid treatment is permitted at doses as per local SoC.For non-COVID-19 disorders, ongoing corticosteroid treatment is permitted at doses up to and including prednisolone 10 mg daily or equivalent.

In patients in the Netherlands only, the use of hydroxychloroquine and/or chloroquine in the past 2 weeks are exclusionary.

* Serum alanine transaminase (ALT) or aspartate transaminase (AST) >5 times upper limit of normal detected within 24 hours at screening or at baseline (according to local laboratory reference ranges) or other evidence if severe hepatic impairment (Child-Pugh Class C).
* Absolute peripheral blood neutrophil count of ≤1000/mm3.
* Estimated GFR (eGFR) ≤30 mL/min/1.73m2 (based on CKD-EPI formula).
* Patients currently being treated with drugs known to be strong or moderate inducers of isoenzyme CYP2C9 and/or strong inhibitors of CYP2C9 and/or strong inducers of cytochrome P450, family 3, subfamily A (CYP3A) and the treatment cannot be discontinued or switched to a different medication prior to starting study treatment.
* Patients with innate or acquired immunodeficiencies.
* Patients who have undergone solid organ or stem cell transplantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Hvidovre, Denmark
- Germany (3):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Budapest, Hungary
- India (3):
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, New Delhi
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico CP
  - Novartis Investigative Site, Monterrey, Nuevo León
- Novartis Investigative Site, Harderwijk, Netherlands
- Peru (2):
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
- Russia (7):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, George, Western Cape, South Africa
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Madurka I, Vishnevsky A, Soriano JB, Gans SJ, Ore DJS, Rendon A, Ulrik CS, Bhatnagar S, Krishnamurthy S, Mc Harry K, Welte T, Fernandez AA, Mehes B, Meiser K, Gatlik E, Sommer U, Junge G, Rezende E; Study group. DFV890: a new oral NLRP3 inhibitor-tested in an early phase 2a randomised clinical trial in patients with COVID-19 pneumonia and impaired respiratory function. Infection. 2023 Jun;51(3):641-654. doi: 10.1007/s15010-022-01904-w. Epub 2022 Sep 14. PMID 36104613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 30 sites in 12 countries.
Pre-assignment Details: Participants underwent a Screening period of up to 24 hours which included screening and baseline assessments.
Period: Overall Study
Arm/Group | DFV890 + SoC | Standard of Care (SoC)
Started (All randomized Participants) | 71 | 72
Safety Analysis Set (All randomized participants, who attended at least one post-baseline visit) | 70 (One participant that was randomized to the DFV890 + SoC arm did not attend any post-baseline visit) | 72
PD Analysis Set (All randomized participants with no protocol deviations with relevant impact on Pharmacodynamics (PD) data) | 62 | 68
Completed | 62 | 59
Not Completed | 9 | 13
Not completed — Death | 6 | 8
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Deviation | 1 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DFV890 + SoC | Standard of Care (SoC) | Total
Number analyzed (Participants) | 71 | 72 | 143
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (13.31) | 61.5 (10.38) | 60.8 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 49 | 48 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 5 | 11
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 55 | 57 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: APACHE II Severity of Disease Score on Day 15 or on the Day of Discharge (Whichever is Earlier)
Description: The APACHE II ("Acute Physiology And Chronic Health Evaluation II") is a severity-of-disease classification system. An integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death. In practice, it is rare for any participant to accumulate more than 55 points.
  APACHE II score was measured on Day 15 or on the day of discharge (whichever was earlier). Participants who died on Day 15 or earlier were assigned the highest observed APACHE II score of any of the participants at any time during the trial (worst case imputation for deaths). Missing data values of the parameters required for the derivation of the APACHE II score were replaced by the last available assessment.
Time Frame: up to Day 15
Population: Safety analysis set: All randomized participants, who attended at least one post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | DFV890 + SoC | Standard of Care (SoC)
Number analyzed (Participants) | 70 | 72
Score on a scale | 8.7 (1.06) | 8.6 (1.05)
Statistical Analysis 1: Comparison: DFV890 + SoC vs Standard of Care (SoC); Test type: Superiority; p = 0.467, ANCOVA; Least squares mean difference = 0.11, 90% CI 2-sided [-2.0 to 2.3], Standard Error of Mean 1.297

2. Secondary Outcome: Serum C-reactive Protein (CRP) Levels
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. It was analyzed on a log-scale fitting a repeated measures mixed model including treatment group, study day, the three stratification factors and log transformed baseline CRP as a covariate. Values reported were back-transformed to original scale.
Time Frame: Days 2, 4, 6, 8, 10, 12, 14 and 15
Population: PD analysis set: All randomized participants with no protocol deviations with relevant impact on PD data.
Measure: Geometric Mean (Standard Error); unit: Milligram / Liter
Arm/Group | DFV890 + SoC | Standard of Care (SoC)
Number analyzed (Participants) | 62 | 68
Milligram / Liter
  Day 2: number analyzed (Participants) | 60 | 66
  Day 2 | 31.4 (1.14) | 46.6 (1.13)
  Day 4: number analyzed (Participants) | 57 | 61
  Day 4 | 22.2 (1.19) | 26.5 (1.18)
  Day 6: number analyzed (Participants) | 52 | 60
  Day 6 | 11.5 (1.2) | 15.1 (1.19)
  Day 8: number analyzed (Participants) | 50 | 55
  Day 8 | 7.7 (1.25) | 10.9 (1.24)
  Day 10: number analyzed (Participants) | 41 | 40
  Day 10 | 7.0 (1.27) | 8.0 (1.27)
  Day 12: number analyzed (Participants) | 38 | 28
  Day 12 | 7.5 (1.30) | 7.1 (1.31)
  Day 14: number analyzed (Participants) | 34 | 26
  Day 14 | 8.1 (1.31) | 6.3 (1.31)
  Day 15 / end of study: number analyzed (Participants) | 49 | 51
  Day 15 / end of study | 6.9 (1.27) | 8.2 (1.26)
Statistical Analysis 1: Comparison: DFV890 + SoC vs Standard of Care (SoC); Test type: Superiority; p = 0.237, Mixed Models Analysis — One-sided; p-value reported is for the treatment factor across all time points

3. Secondary Outcome: Clinical Status Over Time
Description: Clinical status was measured with World Health Organization (WHO) 9-point ordinal scale.
  The scoring is - Uninfected patients have a score 0. - Ambulatory patients can have a score 1 (no limitation of activities) or 2 (limitation of activities). - Hospitalized patients with mild disease can have score 3 (no oxygen therapy) or 4 (oxygen by mask or nasal prongs). - Hospitalized patients with severe disease can have score 5 (non-invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support - pressors, renal replacement therapy, extracorporeal membrane oxygenation). - Patients who die have a score 8.
  Missing data values were handled as follows: For participants who died prior to Day 29, the score for death was imputed for all following visits up to and including day 29. For all the other participants, last observation carried forward was applied up to and including Day 29.
Time Frame: Baseline, days 2, 4, 6, 8, 10, 12, 14, 15, 17, 19, 21, 23, 25, 27 and 29
Population: Safety analysis set: All randomized participants, who attended at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | DFV890 + SoC | Standard of Care (SoC)
Number analyzed (Participants) | 70 | 72
Score on a scale
  Baseline | 4.3 (0.49) | 4.3 (0.44)
  Day 2 | 4.3 (0.58) | 4.3 (0.80)
  Day 4 | 4.3 (0.83) | 4.3 (0.95)
  Day 6 | 3.9 (1.11) | 4.2 (1.13)
  Day 8 | 3.8 (1.31) | 3.8 (1.50)
  Day 10 | 3.6 (1.48) | 3.6 (1.88)
  Day 12 | 3.4 (1.66) | 3.3 (1.98)
  Day 14 | 3.3 (1.75) | 3.1 (2.03)
  Day 15 | 2.8 (2.02) | 2.6 (2.24)
  Day 17 | 2.7 (2.01) | 2.5 (2.22)
  Day 19 | 2.6 (2.01) | 2.5 (2.27)
  Day 21 | 2.6 (2.01) | 2.5 (2.33)
  Day 23 | 2.6 (2.03) | 2.4 (2.31)
  Day 25 | 2.6 (2.07) | 2.4 (2.31)
  Dy 27 | 2.6 (2.10) | 2.4 (2.31)
  Day 29 | 1.9 (2.34) | 1.9 (2.57)

4. Secondary Outcome: Number of Participants Not Requiring Mechanical Ventilation for Survival
Description: Number of participants not requiring mechanical ventilation for survival until Day 15 and Day 29: defined by WHO 9-point ordinal scale score of < 6 points at all time points assessments.
  The scoring is - Uninfected patients have a score 0. - Ambulatory patients can have a score 1 (no limitation of activities) or 2 (limitation of activities). - Hospitalized patients with mild disease can have score 3 (no oxygen therapy) or 4 (oxygen by mask or nasal prongs). - Hospitalized patients with severe disease can have score 5 (non-invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support). - Patients who die have a score 8.
  Missing data values were handled as follows: For participants who died prior to Day 29, the score for death was imputed for all following visits up to and including day 29. For all the other participants, last observation carried forward was applied up to and including Day 29.
Time Frame: Until Day 15 (Assessments on Days 2, 4, 6, 8, 10, 12, 14 and 15) and until Day 29 (Assessments on Days 17, 19, 21, 23, 25, 27 and 29)
Population: Safety analysis set: All randomized participants, who attended at least one post-baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | DFV890 + SoC | Standard of Care (SoC)
Number analyzed (Participants) | 70 | 72
Participants
  Until Day 15 | 60 | 59
  Until Day 29 | 60 | 58

5. Secondary Outcome: Number of Participants With at Least One-point Improvement From Baseline in Clinical Status
Description: Number of participants with at least one-point improvement from baseline in clinical status, which was measured with WHO 9-point ordinal scale.
  The scoring is - Uninfected patients have a score 0. - Ambulatory patients can have a score 1 (no limitation of activities) or 2 (limitation of activities). - Hospitalized patients with mild disease can have score 3 (no oxygen therapy) or 4 (oxygen by mask or nasal prongs). - Hospitalized patients with severe disease can have score 5 (non-invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support). - Patients who die have a score 8.
  Missing data values were handled as follows: For participants who died prior to Day 29, the score for death was imputed for all following visits up to and including day 29. For all the other participants, last observation carried forward was applied up to and including Day 29.
Time Frame: Baseline, Day 15 and Day 29
Population: Safety analysis set: All randomized participants, who attended at least one post-baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | DFV890 + SoC | Standard of Care (SoC)
Number analyzed (Participants) | 70 | 72
Participants
  Day 15 | 59 | 53
  Day 29 | 61 | 60

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start of treatment to 30 days after end of treatment, assessed up to maximum duration of 45 days.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- Total: Total
Arm/Group | DFV890 + SoC | Standard of Care (SoC) | Total
All-Cause Mortality (participants affected / at risk) | 8/70 | 8/72 | 16/142
Serious Adverse Events (participants affected / at risk) | 16/70 | 11/72 | 27/142
Other Adverse Events (participants affected / at risk) | 12/70 | 6/72 | 18/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DFV890 + SoC (N=70) | Standard of Care (SoC) (N=72) | Total (N=142)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Condition aggravated (General disorders) | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 2 | 4
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 2 | 3
Septic shock (Infections and infestations) | 1 | 1 | 2
Amylase increased (Investigations) | 1 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 8
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 1
Haemodynamic instability (Vascular disorders) | 0 | 2 | 2
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DFV890 + SoC (N=70) | Standard of Care (SoC) (N=72) | Total (N=142)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 10
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT04382053/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT04382053/SAP_001.pdf